CLINICAL TRIAL: NCT00974831
Title: Glucose Tolerance in Healthy Overweight Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Bobbie L Swearengin, RN, Abbott Nutrition
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BK51
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AA Drink (Experimental): Amino Acid Drink Mixture
  Interventions: Other: Amino Acid Drink Mixture
- Glucose drink (Placebo Comparator)
  Interventions: Other: Glucose drink

INTERVENTIONS:
Other: Amino Acid Drink Mixture — 22 oz consumed in 7 oz, 8oz, 7 oz increments 5 minutes apart over 15 mins
  Arms: AA Drink
Other: Glucose drink — 22 oz consumed in 7 oz, 8oz, 7 oz increments 5 minutes apart over 15 mins
  Arms: Glucose drink

SUMMARY:
The primary objective is to compare the postprandial glycemic response of healthy overweight adults after consuming an amino acid drink mix versus a control drink.

ELIGIBILITY:
Inclusion Criteria:

1. Fasting blood glucose level of ≥ 70mg/dL and ≤ 125 mg/dL.
2. Subject states that he/she does not have type 1 or 2 diabetes.
3. Subject is overweight as defined as waist circumference ≥ 101 cm (40 inches) male; ≥ 88 cm (35 inches) female.
4. Subject's BMI is ≥ 25 kg/m2.
5. Subject's blood pressure is < 140 mm Hg systolic and < 90 mm Hg diastolic.
6. Subject is between 20 and 45 years of age, inclusive.
7. Subject is a male or a non-pregnant, non-lactating female, at least 6 weeks postpartum prior to screening visit.
8. If female is of childbearing potential, is practicing birth control
9. If subject is on a chronic medication such as a thyroid medication or hormone therapy, has been on constant dosage for at least two months prior to screening visit.

Exclusion Criteria:

1. Subject is eating a low carbohydrate diet such as Atkins, Zone, or South Beach diet plan.
2. Subject states that he/she has current infection, has had inpatient surgery, or corticosteroid treatment in the last 3 months or antibiotics in the last 3 weeks prior to screening visit.
3. Subject states that he/she has an active malignancy.
4. Subject states that he/she has had a significant cardiovascular event ≤ six months prior to screening visit; or stated history of congestive heart failure.
5. Subject states that he/she has end-stage organ failure or is status post organ transplant.
6. Subject states that he/she has a history of renal disease.
7. Subject states that he/she has current hepatic disease.
8. Subject states that he/she has a chronic, contagious, infectious disease, such as active tuberculosis, Hepatitis B or C, or HIV.
9. Subject has taken/is currently taking any herbals, dietary supplements, or medications during the past four weeks prior to screening visit that could profoundly affect blood glucose.
10. Subject has taken/is currently taking any herbals, dietary supplements, or medications during the past four weeks prior to screening visit to control hypertension or cholesterol.
11. Subject states that he/she has clotting or bleeding disorders.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The primary variable is the positive area under the curve from 0 to 180 minutes for plasma glucose. | 0-180 minutes

SECONDARY OUTCOMES:
Plasma glucose, insulin, C-peptide, free fatty acids, and glucagon concentration data over time | 0-180 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Nelson, PhD, Study Chair — Abbott Nutrition
Locations (1):
- University of Texas, Austin, Texas, United States